CLINICAL TRIAL: NCT02950857
Title: A Phase Ib, Open-label, Repeat Dose, Study of EPEG in Beta Thalassemia Patients With Non-transfusion Dependent Thalassemia (β NTDT)
Brief Title: A Study of EPEG in Beta Thalassemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETH-001
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPEG (pegylated erythropoietin) - 0.9 µg/kg (Experimental): Four weekly subcutaneous injections of 0.9 µg/kg EPEG
  Interventions: Drug: EPEG
- EPEG (pegylated erythropoietin) - 1.2 µg/kg (Experimental): Four weekly subcutaneous injections of 1.2 µg/kg EPEG
  Interventions: Drug: EPEG
- EPEG (pegylated erythropoietin) - 1.5 µg/kg (Experimental): Four weekly subcutaneous injections of 1.5 µg/kg EPEG
  Interventions: Drug: EPEG

INTERVENTIONS:
Drug: EPEG — (Pegylated erythropoeitin)

SUMMARY:
An open-label study in which 6 patients will receive once-weekly subcutaneous injections of EPEG for 4 weeks. Final visit will occur 60 days after study entry

DETAILED DESCRIPTION:
Following the provision of informed consent, screening visit procedures to be performed will include: a detailed medical history (including concomitant medications), physical exam, vital signs (non-invasive systolic and diastolic arterial blood pressure, heart rate, and respiratory rate, temperature, and oxygen saturation by pulse oximetry,), laboratory testing of blood samples collections for safety (hematology and chemistry), and urinalysis (dipstick and microscopy, if necessary). A serum pregnancy test for all female patients (of child-bearing potential) will be measured during the Screening Visit. Urine pregnancy test for all female patients (of child-bearing potential) will be measured at each dosing visit prior to dosing.

Eligible patients will receive either subcutaneous injection of EPEG (0.9 µg/kg, 1.2 µg/kg, and 1.5 µg/kg,) for four weeks followed by follow up for 5-6 weeks after 4th dose of IP.

Vital signs will be recorded for study documentation at 1 hour after dosing and at discharge of the day (to occur 2 hours after the time of dosing). All patients will receive standard of care as per investigative site standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 - 65 years of age
3. Confirmed diagnosis of Non-Transfusion Dependent β-thalassemia (β-NTDT)
4. Hemoglobin 6.0-10.0 g/dL
5. Signed and dated informed written consent by the subject
6. Able to receive subcutaneous injections of study drug
7. Female patients must be non-lactating
8. Female patients of reproductive potential must have a negative serum pregnancy (β-HCG) test at screening.

Exclusion Criteria:

1. In the judgment of the investigator the patient is not a good candidate for the study
2. Blood transfusion within the last 30 days
3. Any of the following medical conditions:

   1. Severe kidney insufficiency, defined as use of hemodialysis or serum creatinine at levels greater than 2.5 mg/dL at the time of screening
   2. Cardiac disease with adjustment of cardiac medications in the 60 days before study entry
   3. Symptomatic coronary artery disease, as indicated by a history of chest pain, angina, claudication, or surgery to treat coronary artery disease in the 1 year before study entry
   4. Stroke, defined as a new focal neurological deficit lasting more than 24 hours in the 45 days before study entry
   5. New diagnosis of pulmonary embolism by ventilation-perfusion scan, angiography, or any other technique in the 90 days before study entry
   6. History of retinal detachment or retinal hemorrhage in the 180 days before study entry
   7. Use of nitrate-based vasodilators, prostacyclin (inhaled, subcutaneous, or intravenous)
   8. Acute asthma exacerbation requiring use of prednisone in the 60 days before study entry
   9. Initiation or dosage increase of calcium channel blockers in the 30 days before study entry
   10. Initiation of any other cardiac or pulmonary medication in the 90 days before study entry
4. Presence of any other condition, which in the opinion of the investigator, would make the person unsuitable for enrollment or could interfere with compliance in the study, including but not limited to alcohol or drug abuse
5. Any prior treatment with Erythropoiesis-stimulating Agents (ESA) within 90 days of study treatment;
6. History of hypersensitivity to erythropoietin or any related drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Number of participants in each treatment arm with abnormal laboratory values and/or adverse events that are related to treatment. | 60 days
  Safety of treatment as determined by changes in vital signs, chest X-Ray, electrocardiographic, biochemical, hematological, and urinalysis measures, and reported adverse events

SECONDARY OUTCOMES:
Change in the Hemoglobin from Baseline to the Final Visit | 60 Days
A mean increase in Hematocrit (Hct) from Baseline to the Final Visit | 60 Days
A mean increase in reticulocyte count from Baseline to the Final Visit | 60 Days
Change in clinical signs and symptoms of β-NTDT from Baseline to the Final Visit | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Real, MD, Study Director — Prolong Pharmaceuticals
Locations (1):
- Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No